CLINICAL TRIAL: NCT07141121
Title: Feasibility of Timesaving When Using Histolog Confocal Laser Endomicroscopy for Margin Assessment in Prostatectomy Specimen
Acronym: IMARHGIN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: SamanTree Medical SA (Industry)
Responsible Party: Principal Investigator, Ashutosh Kumar Tewari, Professor and System Chairman, Department of Urology, Icahn School of Medicine at Mount Sinai
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: STUDY-24-01611
Record Dates: First submitted 2025-07-31; First posted 2025-08-26 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-10

CONDITIONS: Prostate Cancer
Keywords: Confocal Microscopy; Histolog Scanner; NeuroSafe; Surgical Margins; Feasibility; Radical Prostatectomy
MeSH Terms: conditions — Prostatic Neoplasms; Margins of Excision

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Patients undergoing robotic-assisted radical prostatectomy (Experimental): Patients undergo standard of care (SOC) robotic-assisted radical prostatectomy. The patients' removed prostates are then evaluated with the Histolog Scanner. Patients also undergo SOC blood sample collection, rectal examination, MRI, and micro ultrasound imaging, as well as have their medical records reviewed throughout the trial.
  Interventions: Device: Histolog Scan

INTERVENTIONS:
Device: Histolog Scan — Upon prostate removal, the prostate is taken to the Histolog scanner, dipped in proprietary fluorescent dye, rinsed with saline, and then scanned on five different sides. This involves simply placing the prostate on the surface of the scanner and acquiring images on each side, giving a high-resolution (cellular level) microscopic imaging of the prostate's surfaces. Once images are collected, the prostate is returned to the pathology lab to undergo the NeuroSafe procedure, which is standard of care (SOC).

SUMMARY:
This study investigates a new, faster way to find cancer cells on the surface of the prostate during radical prostatectomy surgery. A recently FDA-approved device, called the Histolog Scanner, gives high-resolution imaging of the surface of fresh tissue using ultra-fast confocal microscopy, which allows physicians to make surgical decisions quickly.

DETAILED DESCRIPTION:
The goal of this time saving feasibility study is to gain early insights into whether Histolog Scanner can maintain the integrity and safety of NeuroSafe margin assessment while alleviating the heavy time burden of NeuroSafe in the US setting before starting a larger clinical trial. This way, patients can be offered optimal nerve sparing without adding to the administrative burden and cost associated with NeuroSafe. What is new about the study is that the researchers intend to do a cost and time economics analysis using United States market prices that will inform discussions in the future about the utility of this device in the United States.

ELIGIBILITY:
Inclusion criteria:

* Localized or locally advanced prostate cancer D'Amico intermediate or high-risk disease.
* Indicated for robot-assisted radical prostatectomy
* Treatment naive.
* Age ≥ 18 years.
* Ability to understand and the willingness to sign a written informed consent.

Exclusion criteria:

* Patients who have received pelvic radiation previously for prostate cancer or any other malignancy.
* Patients who have previously received androgen deprivation or other hormonal treatments, or focal therapy of prostate cancer prior to radical prostatectomy.
* Patients with D'Amico Criteria low risk prostate cancer.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — This study is looking at post-surgical specimens for patients with prostate cancer, so the researchers are only looking at a male population.
Enrollment: 78 (Estimated)
Dates: Start 2025-05-13 (Actual); Primary Completion 2026-05-13 (Estimated); Study Completion 2026-05-13 (Estimated)

PRIMARY OUTCOMES:
Proportion of Surgeries with Histolog Scanner Attributable Time-Saving Greater Than 20 Minutes | Immediately after procedure
  Defined as a positive difference of time taken using NeuroSafe technique vs time taken by Histolog scanner in margin assessment.

SECONDARY OUTCOMES:
Agreement Between Histolog and Final Histopathology Assessment | Immediately after procedure
  The Kappa statistic (Cohen's Kappa) will be used to assess agreement between Histolog and final histopathology assessment. 95% CI will be calculated using the Wilson's method without continuity correction.
System Usability Scale (SUS) | "Baseline" or "Day 1" and through study completion, an average of 1 year
  System Usability Scale (SUS) ranges between 8-40. Each question asks about ease of use of the Histolog Scanner, and the operator answers each of the 8 questions on a scale of 1 (strongly disagree) to 5 (strongly agree). Any SUS score greater than or equal to 32 will be interpreted as high usability.
  Operator will be asked to complete after the completion of every 10 procedures and again after the final procedure.
Pathologist Usability Scale (PUS) score | "Baseline" or "Day 1" and through study completion, an average of 1 year
  Pathologist Usability Scale (PUS) ranges between 6-30. Each question asks about the ease of use of the Histolog Scanner, and the pathologist answers each of the 6 questions on a scale of 1 (strongly disagree) to 5 (strongly agree). Any PUS score greater than or equal to 25 will be interpreted as high pathologist usability.
  Pathologist will be asked to complete after the completion of every 10 procedures and again after the final procedure.
Count and percentage of specimens where the Histolog Dip impacted the ability to make final margin assessments in pathology | Immediately after procedure
  Count and percentage of specimens where the Histolog Dip impacted the ability to make final margin assessments in pathology

CONTACTS AND LOCATIONS:
Overall Officials: Ashutosh K. Tewari, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol
Time Frame: Specify Other Time FrameTBD
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee ('learned intermediary') identified for this purpose.
  For individual participant data meta-analysis. Proposals may be submitted up to 36 months following article publication. After 36 months the data will be available in the University's data warehouse but without investigator support other than deposited metadata. Information regarding submitting proposals and accessing data may be found at (to be determined).